CLINICAL TRIAL: NCT03622619
Title: The Effect of Manuka Eye Drops on Tear Film Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Jacqueline Tan-Showyin, Senior Research Fellow, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOVS2018-501
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Manuka eye drops (Experimental)
  Interventions: Other: Optimel Antibacterial Manuka+ Dry Eye Drops
- Systane Ultra (Active Comparator)
  Interventions: Other: Systane Ultra Lubricating Eye Drops

INTERVENTIONS:
Other: Optimel Antibacterial Manuka+ Dry Eye Drops — Leptospermum sp Honey 165mg/g
  Arms: Manuka eye drops
Other: Systane Ultra Lubricating Eye Drops — Polyethylene glycol 400 0.4% and propylene glycol 0.3%
  Arms: Systane Ultra

SUMMARY:
Traditionally, Manuka honey has been used to combat against bacteria and reduce inflammation (the body's way of reacting to infection, irritation or other injury). Due to the inflammatory nature of dry eye, Manuka eye drops show promise as a treatment for dry eye disease. The aim of this research is to compare the effects of two over the counter eye drops that are used to treat dry eye conditions over a one month period.

DETAILED DESCRIPTION:
The aim of the present study is to conduct a randomised clinical trial to compare the effect on tear film properties and dry eye signs and symptoms of Optimel Manuka eye drops compared to Systane Ultra, a widely available over the counter aqueous tear supplement as a control eye drop. This investigation will involve a minimum of 40 participants who have dry eye, who are randomly put into two groups receiving either Optimel Manuka drops or Systane Ultra used three times daily for one month. Both of these products are commercially available in Australia. Results from this study will inform practitioners as to the potential benefits of Manuka eye drops on tear film characteristics and signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend English and give informed consent as demonstrated by signing a record of informed consent;
* General population aged 18 years and over;
* In good general health;
* Subjectively experiencing dry eye symptoms (e.g. burning, irritation, and discomfort due to dryness of the eye or exposure to wind or sun). Participants will be selected based on a minimum OSDI score of 13 points (1).
* Willing to discontinue CL wear for 1 week before first visit and continue to do so until the conclusion of the study;
* Participant is willing to discontinue their use of any previous conventional dry eye treatment method commenced before the study throughout the study;
* Willing to comply with the dosage and study visit schedule as directed by the investigator;
* No planned changes to diet and willing not to substantially alter their usual diet for the duration of the study, including their typical intake of fish, green tea or oral supplements known to have anti-inflammatory properties;
* Willingness to notify the study investigator if instructed to alter their diet by health/medical practitioner.

Exclusion Criteria:

* Allergy to benzoic acid preservatives;
* Allergy to honey products;
* Active anterior eye disease/ infection, inflammation/allergy that requires ocular medical treatment;
* Eye injury or surgery in the past 6 months including chemical burns, penetrating injuries, traumatic iritis, orbital fractures, laser surgery, strabismus surgery, cataract or any other intraocular surgeries;
* Soft contact lens, rigid gas permeable, orthokeratology lens wearer within one week prior to the study and during the study.
* Use of any of the following medications (including steroids) up to 12 weeks prior to start of the study or during the course of the study:

  * Ocular medication, category S3 and above;
  * Any systemic or topical medications that will affect ocular physiology e.g. anti-acne medications such as Roaccutane and corticosteroid or immunosuppressant medications such as Hydrocortisone, Prednisolone and antihistamine medications such as Claritine;
* Any systemic disease that may affect ocular health e.g. Graves disease, and auto-immune diseases such as ankolysing spondylitis, multiple sclerosis and systemic lupus erythematosis;
* Epilepsy or history of migraines exacerbated by flashing, strobe-like lights.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Tan, PhD, Principal Investigator — University of New South Wales
Locations (1):
- School of Optometry and Vision Science, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Study results will be made available in the form of summaries

REFERENCES:
- [Derived] Tan J, Jia T, Liao R, Stapleton F. Effect of a formulated eye drop with Leptospermum spp honey on tear film properties. Br J Ophthalmol. 2020 Oct;104(10):1373-1377. doi: 10.1136/bjophthalmol-2019-315160. Epub 2020 Jan 16. PMID 31949092

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Manuka Eye Drops | Systane Ultra
Started | 23 | 23
Completed | 21 | 21
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manuka Eye Drops | Systane Ultra | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.20 (3.47) | 20.56 (3.16) | 21.39 (3.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 9 | 5 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian | 17 | 15 | 32
  Ethnicity: Non-Asian | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  Australia | 21 | 21 | 42
Ocular Surface Disease Index Score [Mean (Standard Deviation); unit: scores on a scale] — The Ocular Surface Disease Index (OSDI) dry eye questionnaire evaluated dry eye severity on a scale of 0 to 100, with higher scores representing greater severity of dry eye. Those with an OSDI score of below 13 were excluded.
  scores on a scale | 33.65 (12.38) | 28.17 (12.31) | 30.91 (12.51)

OUTCOME MEASURES:

1. Primary Outcome: A Measurable Difference in Tear Lipid Layer Thickness After 4 Weeks of Daily Use
Description: The primary endpoint is a measurable difference in tear lipid layer thickness between Optimel Manuka eye drops and Systane Ultra eye drops after 4 weeks of daily use. Tear film inferior lipid layer thickness (LLT; nm) is measured using the LipiView II (Johnson and Johnson Vision, USA). The participant's eye is positioned in front of an illumination source that is directed toward the tear film on the corneal surface. The camera records a 20-second video of the tear film interference and subsequently displays a value in interferometric colour units (ICU), where 1 ICU approximates 1nm of lipid layer thickness.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Manuka Eye Drops | Systane Ultra
Number analyzed (Participants) | 21 | 21
nm | -5.1 (22.2) | -3.2 (21.8)
Statistical Analysis 1: Comparison: Manuka Eye Drops vs Systane Ultra; Test type: Other; p = 0.65, Wilcoxon (Mann-Whitney)

2. Primary Outcome: A Measurable Difference in Tear Evaporation Rate After 4 Weeks of Daily Use.
Description: A measurable difference in Tear evaporation rate between Optimel Manuka eye drops and Systane Ultra eye drops after 4 weeks of daily use. Measured using a Modified Vapometer. The Modified Vapometer is a closed chamber device which is used for measuring transepidermal water loss. Participants will be seated upright on a chair and provided with a distance fixation target. To minimize the effect of skin evaporation, petroleum jelly (Vaseline, http://www.unilever.com.au/brands-in-action/detail/Vaseline/299339/) will be applied over the upper eyelid and the surrounding areas. The VapoMeter will then be placed over the eye and a non-invasive measurement of tear evaporation will be taken within 10 s. Participants will be instructed not to blink during open eye measurement and to maintain a normal straight gaze at the fixation target. Evaporation rates with the eyes closed will also be taken, in order to account for the skin evaporation from eyelids and surrounding skin tissue.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: gm-2h
Arm/Group | Manuka Eye Drops | Systane Ultra
Number analyzed (Participants) | 21 | 21
gm-2h | -10.8 (16.7) | 0.7 (10.8)
Statistical Analysis 1: Comparison: Manuka Eye Drops vs Systane Ultra; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney)

3. Primary Outcome: A Measurable Difference in Fluorescein Tear Break-up Time After 4 Weeks of Daily Use
Description: A measurable difference in fluorescein tear break-up time between Optimel Manuka eye drops and Systane Ultra eye drops after 4 weeks of daily use. Fluorescein tear break-up time (TBUT; sec) (Opti-Strip-FL, Optimed, Lane Cove West, NSW, Australia) was measured viewed with a yellow Wratten filter (No. 12, Kodak) and cobalt light of the slit lamp biomicroscope. Three consecutive TBUT measurements for each eye were taken by a single masked investigator.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Manuka Eye Drops | Systane Ultra
Number analyzed (Participants) | 21 | 21
seconds | 2.0 (3.0) | 0.0 (3.1)
Statistical Analysis 1: Comparison: Manuka Eye Drops vs Systane Ultra; Test type: Superiority; p = 0.055, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: A Measurable Difference in Subjective Symptoms After 4 Weeks of Daily Use
Description: A measurable difference in subjective symptoms between Optimel Manuka eye drops and Systane Ultra eye drops after 4 weeks of daily use. Subjective symptoms is measured using an visual analogue scale ranging from 0 to 100, with higher scores meaning worse outcome. Participants are asked to visually represent their symptom severity by marking a dot on a line ten centimetres in length. These are then measured using a ruler to the nearest 0.5mm and given a score from zero to 100, with zero indicative of no symptoms and 100 suggesting maximum symptom severity
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manuka Eye Drops | Systane Ultra
Number analyzed (Participants) | 21 | 21
units on a scale
  Burning/stinging | -10.7 (23.2) | -8.9 (18.6)
  Grittiness/foreign body sensation | -20.8 (20.4) | -15.0 (17.9)
  Dryness | -35.4 (22.1) | -32.2 (19.2)
  Blurry vision | -13.6 (22.5) | -20.6 (29.8)
  Overall discomfort | -14.7 (15.1) | -10.7 (17.5)
Statistical Analysis 1: Comparison: Manuka Eye Drops vs Systane Ultra; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney); Burning/stinging
Statistical Analysis 2: Comparison: Manuka Eye Drops vs Systane Ultra; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney); Grittiness/foreign body sensation
Statistical Analysis 3: Comparison: Manuka Eye Drops vs Systane Ultra; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney) — Dryness
Statistical Analysis 4: Comparison: Manuka Eye Drops vs Systane Ultra; Test type: Superiority; p = 0.14, Wilcoxon (Mann-Whitney) — Blurred vision
Statistical Analysis 5: Comparison: Manuka Eye Drops vs Systane Ultra; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney) — Overall discomfort

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Manuka Eye Drops | Systane Ultra
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manuka Eye Drops (N=21) | Systane Ultra (N=21)
Ocular Stinging (Eye disorders) | 1 (1) | 0 (0) — Stinging sensation of the eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03622619/Prot_SAP_000.pdf